CLINICAL TRIAL: NCT01511068
Title: Inhaled Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in Hereditary Pulmonary Alveolar Proteinosis (PAP)
Acronym: FAMPAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Virginia Commonwealth University (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0959_CCHMC_IRB; NCT01534156 (obsolete NCT alias)
Record Dates: First submitted 2011-12-12; First posted 2012-01-18 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Hereditary Pulmonary Alveolar Proteinosis
Keywords: PAP
MeSH Terms: interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Leukine (rhGM-CSF) (Experimental): Inhaled recombinant human GM-CSF in individuals with hereditary Pulmonary Alveolar Proteinosis (hPAP) due to partial dysfunction of the GM-CSF receptor
  Interventions: Drug: Leukine

INTERVENTIONS:
Drug: Leukine — Participants will receive inhaled rhGM-CSF (Sargramostim, Leukine) at the dose of 250 mcg one time per week for 12 weeks. Following an interim safety evaluation, participants may be entered into a second 12 week treatment period where participants will receive either 250 mcg or 500 mcg once weekly. At the end of any treatment period, participants will be followed for 12 additional weeks in the absence of inhaled rhGM-CSF to evaluate safety and efficacy.
  Other Names: GM-CSF [Leukine (Sargramostim)]

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of inhaled recombinant human GM-CSF in individuals with hereditary Pulmonary Alveolar Proteinosis (PAP) due to partial dysfunction of the GM-CSF receptor.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PAP caused by bi-allelic mutations in CSF2RA or CSF2RB associated with impaired GM-CSF-R-alpha or GM-CSF-R-beta function, respectively, resulting in reduced but non-zero GM-CSF signaling
* Able and willing to give written informed consent / assent as necessary
* Clinically stable

Exclusion Criteria:

* Confirmed diagnosis of a disorder of surfactant production caused by bi-allelic mutations in ABCA3, SFTPB, or SFTPC
* Confirmed diagnosis of autoimmune PAP caused by a high level of GM-CSF autoantibody
* Confirmed diagnosis of secondary PAP caused by an underlying clinical disorder known to be associated with the development of PAP, e.g., inhalation of silica or titanium; myelodysplasia and others
* Treatment with any investigational agent in the 3 months prior to enrollment
* History of severe allergic or anaphylactic reactions to GM-CSF or other yeast-derived products
* History of asthma or other reactive airways disease
* Known active, viral, fungal, mycobacterial, or other infection
* A serious medical condition which, in the opinion of the investigator or data and safety monitoring committee, would make the patient unsuitable for the study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Bruce Rubin, MD, FRCPC, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Leukine (rhGM-CSF)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Time (Minutes) to Discontinuation of Exercise During a Standardized Treadmill Exercise Test
Description: A modified Bruce protocol stress test was used to evaluate improvement in blood oxygen saturation (SpO2). A pulse-oximeter was placed on the participant's finger with the participant at rest while sitting in a chair. Leads for the electrocardiograph were placed on the chest wall. The treadmill was started at 1.7 miles per hour (mph) and a grade of 0%. At three minute intervals, the speed increased as follows: 1.7 mph, 1.7 mph, 1.7 mph, 2.5 mph, 3.4 mph, 4.2 mph, 5.0 mph, 5.5 mph, 6.0 mph, 6.5 mph, 7.0 mph, and 7.5 mph. The participant stopped the test due to intolerable dyspnea or if the SpO2 fell below 88%.
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 | 17
  Participant 2 | 33

2. Secondary Outcome: Change in Diffusion Capacity for Carbon Monoxide
Description: Routine full pulmonary function testing, including spirometry, lung volumes, and DLCO, were performed according to American Thoracic Society guidelines.
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 | 11
  Participant 2 | 4

3. Secondary Outcome: Change in Minimum Pulse Oximetry During a Standardized Exercise Protocol Oximetry
Description: Standardized exercise pulse oximetry (SEPO) was used to measure SpO2 at the participant's home on a weekly basis between clinic visits. Briefly, a pulse-oximeter was placed on the finger with the participant at rest sitting in a chair. Three baseline (resting) readings were taken over a period of 1 minute to measure the SpO2 at rest. The participant then began stepping onto and off of the first step of a staircase in the home while holding onto the handrail for safety. Stepping was started by placing the bottom of one foot onto the stair followed by the other foot and then removal of one foot from the stair to the floor followed by the other foot. This procedure was repeated at a frequency of 1 cycle per second for a total of 5 minutes. The participant's parent assisted by noting the saturation data at 1-minute intervals during the test onto the weekly exercise form in the participant's Diary. The participant's saturation data continued to be recorded for 3 minutes after the test.
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 | 0
  Participant 2 | 50

4. Secondary Outcome: Change in Radiographic Evidence of PAP Lung Disease
Description: High resolution computed tomography (HRCT) scans were performed using an interval technique, a 1 mm slice was obtained every 20 mm. The slice series were placed so that images were obtained from the pulmonary apices to the lung bases with one of the images located at the level of the carina. The CT parameters were performed at full inspiration and required a lower dose than usual clinical CT scans; 1 mm slices at 20 mm intervals,120 kVp, 60 mAs, rotation time 0.5 second. Images were reconstructed with lung and soft tissue reconstruction kernels (B35F and B60F). The primary analysis was performed using the B60F kernel. Images were read and reported according to Radiology Department protocol. The raw data was recorded on a DVD and sent to CCHMC for centralized reading and lung attenuation analysis.
Time Frame: Baseline, 7 months
Measure: Number; unit: Hounsfield Units
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Hounsfield Units
  Participant 1-Right Lung Baseline | -510
  Participant 1- Right Lung End of Treatment | -579
  Participant 1-Left Lung Baseline | -366
  Participant 1-Left Lung End of Treatment | -441
  Participant 2-Right Lung Baseline | -593
  Participant 2-Right Lung End of Treatment | -675
  Participant 2-Left Lung Baseline | -630
  Participant 2-Left Lung End of Treatment | -726

5. Secondary Outcome: Change in Quality of Life
Description: The PedsQL quality of life questionnaire is a modular approach to measure health-related quality of life in healthy children and those with acute and chronic health conditions. It is self-administered and completed in less than 5 minutes. It contains 23 items divided into 4 domains: physical functioning, emotional functioning, social functioning, and school functioning. To reverse score, transform the 0-4 scale items to 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate a better Health-Related Quality of Life.To create the Psychosocial Health Summary Score, the mean is computed as the sum of the items over the number of items answered in the Emotional, Social, and School Functioning Scales. The Physical Health Summary Score is the same as the Physical Functioning Scale Score. To create the Total Scale Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales.
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 -Total Score | 10.7
  Participant 1 - Physical Health Score | 75
  Participant 1 - Psychosocial Score | -5.2
  Participant 1 - Parent Score | 19.6
  Participant 1 - Child Score | 3.1
  Participant 2 - Total Score | 11.7
  Participant 2 - Physical Health Score | 7.4
  Participant 2- Psychosocial Score | 14.5
  Participant 2 - Parent Score | 5.6
  Participant 2 - Child Score | 18.2

6. Secondary Outcome: Change in Dyspnea Symptom Score
Description: The dyspnea visual analogue scales were used by the patient to record the level of dyspnea by a single mark on a linear scale. The dyspnea scale ranged from 0 to 10, with short of breath all the time equal to 0 and never short of breath equal to 10. A higher score indicated a better dyspnea score.
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 | 71
  Participant 2 | 11

7. Secondary Outcome: Change in Serum Anti-GM-CSF Antibodies Levels
Description: Serum GM-CSF autoantibody was measured as follows: microtiter plates were incubated (4°C, overnight) with rhGM-CSF, washed in PBS and Tween-20, and incubated (room temperature (RT), 1 hour) with blocking solution. Serum samples were diluted with dilution buffer and aliquots of diluted serum or standard were pipetted into adjacent microtiter wells, incubated at RT for 40 minutes, and then washed with wash buffer. Horseradish peroxidase-conjugated secondary antibody was diluted with dilution buffer and pipetted into each well. Plates were incubated (RT, 0.5 hour) and then washed with wash buffer. Substrate solution was added to each well, plates were incubated (RT, 15 min), and color development was stopped with sulfuric acid. Absorbance at 450 nm was measured using a Benchmark® ELISA plate reader.
Time Frame: Baseline and monthly up to 7 months
Measure: Number; unit: micrograms/ml
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
micrograms/ml
  Participant 1-Visit 0-Baseline | 0.67
  Participant 1-Visit 1-Begin Low Dose Therapy | 0.36
  Participant 1-Visit 2 | 0.32
  Participant 1-Visit 3 | 1.85
  Participant 1-Visit 4 | 19.7
  Participant 1-Visit 5-Begin High Dose Therapy | 71.8
  Participant 1-Visit 6 | 118.1
  Participant 1-Visit 7 | 128.2
  Participant 1-Visit 8 - End of Therapy | 110.7
  Participant 2-Baseline | 0.551
  Participant 2-Begin Therapy | 0.358
  Participant 2-Visit 2 | 0.299
  Participant 2-Visit 3 | 81.04
  Participant 2-Visit 4 | 132.52
  Participant 2-Visit 5-Begin High Dose Therapy | 123.66
  Participant 2-Visit 6 | 116.82
  Participant 2-Visit 7 | 104.36
  Participant 2-Visit 8 - End of Therapy | 91.92

8. Primary Outcome: Change in Minimum Pulse Oximetry During a Standardized Treadmill Exercise Test
Description: as for outcome 1
Time Frame: Baseline, 7 months
Measure: Number; unit: Percent Change
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
Percent Change
  Participant 1 | 0
  Participant 2 | -2.1

9. Secondary Outcome: Change in Serum Biomarkers - GM-CSF
Description: Serum GM-CSF was measured via a commercial ELISA kit from R & D Systems.
Time Frame: Baseline and monthly up to 7 months
Measure: Number; unit: picograms/ml
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
picograms/ml
  Participant 1-Visit 0-Baseline | 43.75
  Participant 1-Visit 1-Begin Low Dose Therapy | 39.4
  Participant 1-Visit 2 | 43.2
  Participant 1-Visit 3 | 88.5
  Participant 1-Visit 4 | 11.5
  Participant 1-Visit 5-Begin High Dose Therapy | 7.8
  Participant 1-Visit 6 | 7.8
  Participant 1-Visit 7 | 7.8
  Participant 1-Visit 8 - End of Therapy | 7.8
  Participant 2-Baseline | 26.8
  Participant 2-Begin Therapy | 27.9
  Participant 2-Visit 2 | 24.8
  Participant 2-Visit 3 | 7.8
  Participant 2-Visit 4 | 7.8
  Participant 2-Visit 5-Begin High Dose Therapy | 7.8
  Participant 2-Visit 6 | 7.8
  Participant 2-Visit 7 | 7.8
  Participant 2-Visit 8 - End of Therapy | 7.8

10. Secondary Outcome: Change in Serum Biomarkers - Surfactant Protein D
Description: Surfactant protein D (SP-D) was measured via a commercial ELISA kit from Biovender.
Time Frame: Baseline and monthly up to 7 months
Measure: Number; unit: nanograms/ml
Arm/Group | Inhaled Leukine (rhGM-CSF)
Number analyzed (Participants) | 2
nanograms/ml
  Participant 1-Visit 0-Baseline | 796.2
  Participant 1-Visit 1-Begin Low Dose Therapy | 619
  Participant 1-Visit 2 | 696.4
  Participant 1-Visit 3 | 589
  Participant 1-Visit 4 | 697.2
  Participant 1-Visit 5-Begin High Dose Therapy | 536.9
  Participant 1-Visit 6 | 642.4
  Participant 1-Visit 7 | 495.9
  Participant 1-Visit 8 - End of Therapy | 673.2
  Participant 2-Baseline | 618.7
  Participant 2-Begin Therapy | 469.6
  Participant 2-Visit 2 | 425.5
  Participant 2-Visit 3 | 381.3
  Participant 2-Visit 4 | 401.1
  Participant 2-Visit 5-Begin High Dose Therapy | 298.2
  Participant 2-Visit 6 | 422
  Participant 2-Visit 7 | 456.8
  Participant 2-Visit 8 - End of Therapy | 593

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until the of completion of the study, approximately 1 year.
Arm/Group | Inhaled Leukine (rhGM-CSF)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Leukine (rhGM-CSF) (N=2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Noseblood (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No